CLINICAL TRIAL: NCT07284342
Title: Observational Study Evaluating Subcutaneous LDp/CDp Solution for Infusion Effectiveness on Sleep Disturbances in Advanced Parkinson's Disease
Brief Title: A Study to Assess Change in Sleep Disturbances of Adult Participants With Advanced Parkinson's Disease Receiving Subcutaneous Foslevodopa/Foscarbidopa
Acronym: ONIROS
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-423
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Parkinson's Disease
Keywords: Advanced Parkinson's Disease; Foslevodopa/Foscarbidopa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Foslevodopa/Foscarbidopa: Participants will receive Foslevodopa/Foscarbidopa as prescribed by their physician according to local label.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study will assess change in sleep disturbances of adult participants with advanced Parkinson's disease receiving subcutaneous Foslevodopa/Foscarbidopa under routine clinical practice.

Foslevodopa/Foscarbidopa is an approved drug for the treatment of Parkinson's Disease. Approximately 103 adult participants who are prescribed Foslevodopa/Foscarbidopa by their doctors will be enrolled across approximately 20 sites across Spain.

Participants will receive Foslevodopa/Foscarbidopa subcutaneous infusion as prescribed by their physician. Participants will be followed for up to 12 weekss.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age >=18 years) Advance Parkinson's Disease (aPD) participants, diagnosed of levodopa-responsive idiopathic Symptoms PD (PD) prescribed on foslevodopa/foscarbidopa (LDp/CDp) Subcutaneous solution for infusion (SI) in routine clinical practice following approved Summary of product characteristics (SmPC) (levodopa-responsive Parkinson's disease with severe motor fluctuations and hyperkinesia or dyskinesia when available combinations of Parkinson medicinal products have not given satisfactory results).
* MMSE>=24 (cognitive cut point for the subjects to be able to comply with study procedures).
* Decision to treat with LDp/CDp SI made by the clinician prior to any decision to approach the subject to participate in this study.
* Particpants with moderate to severe obstructive sleep apnea (OSA) (Apnea-Hypoapnea Index (AHI)>15) may be eligible if they comply with treatment (Continuous Positive Airway Pressure (CPAP) device used at least 4 hours/night and 70% of the nights during last month or mandibular advancement device (MAD)) and have an AHI <15.

Exclusion Criteria:

* Participants presenting with contraindications as per LDp/CDp SI SmPC. 2.
* Participants participating in interventional research (not including non-interventional study, Post Marketing Observational Studies (PMOS), or registry participation) at time of enrollment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with advanced Parkinson's disease receiving subcutaneous infusion of Foslevodopa/Foscarbidopa as prescribed by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on Parkinson's Disease (PD)-related sleep disturbances in Advance Parkinson's Disease (aPD) Participants, as assessed by the Parkinson's Disease Sleep Scale - 2 (PDSS-2) | Up to approximately 12 weeks
  The Parkinson's Disease Sleep Scale (PDSS-2) is a self-administered questionnaire and consists of 15 questions on sleep and nocturnal disturbances which can be related to PD. Participants rate each question using a frequency score, ranging from 0 (never) to 4 (very often), the PDSS-2 total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- Spain (13):
  - Hospital Regional Universitario de Malaga /ID# 276357, Málaga, Andalusia
  - Hospital Universitario Marques de Valdecilla /ID# 276315, Santander, Cantabria
  - Hospital General Universitario Santa Lucía /ID# 277222, Cartagena, Murcia
  - Hospital de Cabueñes /ID# 276314, Gijón, Principality of Asturias
  - Hospital Universitario Virgen del Rocio /ID# 277806, Seville, Sevilla
  - Hospital Universitario Torrecárdenas /ID# 276899, Almería
  - Hospital Universitario Vall de Hebron /ID# 276318, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 276319, Barcelona
  - Hospital Universitario De Burgos /ID# 276317, Burgos
  - Hospital Universitario Virgen de las Nieves /ID# 276350, Granada
  - Hospital Universitario Clinico San Cecilio /ID# 276356, Granada
  - Complejo Hospitalario Universitario de Pontevedra /ID# 276313, Pontevedra
  - Hospital Universitario De Toledo /ID# 276884, Toledo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-423